CLINICAL TRIAL: NCT03451409
Title: Neurobiology of Sensory Phenomena in Obsessive-Compulsive Disorder
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-01606
Record Dates: First submitted 2018-01-10; First posted 2018-03-01 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OCD Proband: Healthy controls (HC, n=50) without a family history of OCD will be matched to SIB.
  Interventions: Other: Tasked based functional MRI (fMRI); Other: Eye Tracking Device
- OCD Siblings: Healthy controls (HC, n=50) without a family history of OCD will be matched to SIB.
  Interventions: Other: Tasked based functional MRI (fMRI); Other: Eye Tracking Device
- Healthy Controls: Healthy controls (HC, n=50) without a family history of OCD will be matched to SIB.
  Interventions: Other: Tasked based functional MRI (fMRI); Other: Eye Tracking Device

INTERVENTIONS:
Other: Tasked based functional MRI (fMRI) — 2-3 brief computer tasks while brain activity is being measured. The tasks performed will involve making button press responses to letters, numbers or shapes on the computer screen.
Other: Eye Tracking Device — Camera aimed at eyes to record eye movements during tasks

SUMMARY:
The Research Domain Criteria (RDoC) approach seeks to address the neurobiological mechanisms of sensory symptoms in patients with obsessive-compulsive disorder (OCD) by investigating dimensional components of behavior that more closely align with brain circuitry. This project focuses on the dimensional symptom of sensory phenomena (SP), which are uncomfortable or aversive sensory experiences that drive repetitive behaviors in OCD, including "not just right" sensations, physical urges, and sensations of disgust. SP are very prevalent, occurring in 60-80% of OCD patients, and experienced as highly distressing. Unfortunately, SP are not well addressed by standard treatment approaches, which may be in part because their neurobiological mechanisms are not well understood.

This project builds on our preliminary data to (1) investigate the neural mechanisms of SP in large OCD cohort showing the full range of SP severity and (2) probe for familial risk markers in unaffected siblings of patients. For Aim 1, SP will be measured in 100 OCD patients using the Sensory Phenomena Scale. Diffusion and fMRI data will be acquired during rest and fMRI tasks. In order to identify familial risk markers, Aim 2 will compare sensory phenomena and neural circuitry between OCD probands, 50 unaffected biological siblings of OCD patients, and 50 unrelated healthy controls without a family history of Axis 1 disorders.

DETAILED DESCRIPTION:
This project investigates the neurobiological mechanisms of sensory symptoms in patients with obsessive-compulsive disorder (OCD) and their siblings using task-based fMRI, resting-state functional connectivity, and diffusion MRI approaches. OCD is a chronic disorder presenting a high public health burden. Treatment presents a particular challenge because OCD is extremely heterogeneous, with clusters of symptoms likely derived from differing neural etiologies.

ELIGIBILITY:
Inclusion Criteria:

* Fluent (speaking and writing) in English

Additional criteria for healthy controls (HC):

* Lifetime absence of major Axis I diagnosis according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria
* Not taking psychotropic medications
* No first-degree biological relatives with OCD

Additional criteria for siblings (SIB):

* First-degree biological sibling of a person with OCD

Additional criteria for OCD patients:

* Diagnosis of OCD according to DSM-5 criteria.

Exclusion Criteria:

* Current moderate or high suicidality as assessed through the Mini International Neuropsychiatric Interview (MINI) 7.0.2 suicidality module
* MRI contraindications such as claustrophobia, ferrous implants, braces, or pacemakers
* Major neurological illness (e.g., self-reported history of organic mental syndromes, head trauma, migraines, seizures, other Central Nervous System (CNS) disease, or other significant medical illness that would make participation unsafe or unfeasible)
* Positive urine toxicology or pregnancy test
* Any disability or health problem that prevents them from completing study procedures (e.g. back problems, severe carpal tunnel syndrome, impaired vision that is not corrected with glasses or contact lenses, etc.).
* Present diagnosis of alcohol use disorder or substance use disorder (moderate or severe)
* Present or previous diagnosis of psychosis, bipolar disorder, or major developmental disorder (autism spectrum disorder, intellectual developmental disorder) based on DSM-5 criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will involve 18-60 year-old male or female volunteer subjects of any racial or ethnic group. This will include 100 OCD patients, 50 unaffected biological siblings (SIB) and 50 healthy controls (HC).
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Brain activation in relation to sensory phenomena severity in patients with OCD | 4 Hours
  Statistical modeling using path analysis will test whether brain activation, functional connectivity, and diffusion measures predict Sensory Phenomena (SP) better than alternative models of predictive influence.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Stern, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States